CLINICAL TRIAL: NCT06604442
Title: Intrapatient Comparison of Urinary Radioactivity Following Piflufolastat (18F) and Flotufolastat (18F) PET in Men With Low PSA Biochemical Recurrence of Prostate Cancer Following Radical Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Collaborators: Aixial Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-PSMA-411
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Positron Emission Tomography (PET) Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- piflufolastat (18F) and flotufolastat (18F) positron emission tomography (PET) (Experimental): Each patient will be administered a single dose of piflufolastat (18F) on Day 1, followed by a PET scan. At least 24 hours after the piflufolastat (18F) scan, but within 10 calendar days, all patients will be administered a single dose of flotufolastat (18F) followed by a PET scan.
  Interventions: Drug: Flotufolastat (18F); Drug: piflufolastat (18F)

INTERVENTIONS:
Drug: Flotufolastat (18F) — Positron emission tomography (PET)
Drug: piflufolastat (18F) — Positron emission tomography (PET)

SUMMARY:
Intrapatient Comparison of Urinary Radioactivity Following Piflufolastat (18F) and Flotufolastat (18F) PET in Men with Low PSA Biochemical Recurrence of Prostate Cancer Following Radical Prostatectomy

DETAILED DESCRIPTION:
This is a multi-center, prospective intra-patient comparator study of urinary radioactivity (standardized uptake values [SUV]) following both piflufolastat (18F) and flotufolastat (18F) positron emission tomography (PET) in patients with low prostate-specific antigen (PSA; ≤0.5 ng/mL) biochemical recurrence (BCR) of prostate cancer following radical prostatectomy (RP).

ELIGIBILITY:
Inclusion Criteria:

* Male ≥18 years of age at Visit 1 (Screening).
* Documented history of localized adenocarcinoma of the prostate with prior curative intent treatment with RP and undetectable PSA post-surgery, experiencing BCR of prostate cancer.
* At least 6 months must have elapsed after RP.
* Low PSA BCR defined as PSA ≤0.5 ng/mL.
* Scheduled by their treating physician to receive a PSMA (18F) PET scan.
* Written informed consent obtained from the patient and ability for the patient to comply with the requirements of the study.

Exclusion Criteria:

* Patients with any medical condition or circumstance (including receiving an IP) that the investigator believes may compromise the data collected or lead to a failure to fulfill the study requirements.
* Patients who are planned to have an x-ray contrast agent or any other PET radiotracer within 24 hours prior to either PSMA PET scan.
* Patients who have already received a piflufolastat (18F) PET scan prior to providing informed consent for this study.
* Patients participating in an interventional clinical trial within 30 days and having received an IP within five biological half-lives prior to either of the PSMA PET scans in this study.
* Patients with known hypersensitivity to the active substance or to any of the excipients of piflufolastat (18F) or flotufolastat (18F).
* Patients who have previously undergone a cystectomy or have renal failure, or have other conditions that may significantly affect urinary output, as judged by the investigator.
* Patients who have already received salvage therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
To compare urinary bladder radioactivity observed on piflufolastat (18F) PET and flotufolastat (18F) PET. | Screening, piflufolastat (18F) on Day 1, At least 24 hours after the piflufolastat (18F) scan, but within 10 calendar days
  Difference in urinary bladder mean SUV (SUVmean) between piflufolastat (18F) and flotufolastat (18F).

SECONDARY OUTCOMES:
To assess the following for piflufolastat (18F) PET and flotufolastat (18F) PET: Detection rates; Detection rates stratified by PSA level; Prostate bed detection rates: local recurrences by subregion; Pelvic lymph node (PLN) detection rates | Screening, piflufolastat (18F) on Day 1, At least 24 hours after the piflufolastat (18F) scan, but within 10 calendar days
  Estimate of the following for each radiopharmaceutical: Patient-level detection rate; Patient-level detection rate by baseline PSA categories; Detection rate for local recurrences in prostate bed for the following subregions: vesicourethral anastomosis lesions; retrovesical lesions; remnant seminal vesicles/lateral surgical margin lesions; Detection rate for PLN lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Helfand, M.D., Principal Investigator — Endeavor Health NorthShore Hospital
Locations (9):
- United States (9):
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope Medical Center, Duarte, California
  - Tower Urology, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Endeavor Health- Glenbrook Hospital, Glenview, Illinois
  - XCancer Omaha/Urology Cancer Center, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Urology San Antonio, San Antonio, Texas